CLINICAL TRIAL: NCT05303285
Title: A Multicenter Study Evaluating the Efficacy and Safety of Secukinumab 300mg in Chinese Adults With Active Ankylosing Spondylitis.
Brief Title: A Study Evaluating the Efficacy of Secukinumab 300mg in Chinese Adults With Active Ankylosing Spondylitis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Collaborators: Wuhan Central Hospital (Other); Wuhan Hospital of Traditional Chinese Medicine (Other); Novartis (Industry); Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Principal Investigator, YIKAI YU, Clinical Professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Tongji0228
Record Dates: First submitted 2022-03-08; First posted 2022-03-31 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Ankylosing Spondylitis (AS)
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — secukinumab

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Secukinumab 300mg (Experimental): Induction with secukinumab 150 mg s.c. once per week (Week 0, 1, 2, 3 and 4) followed by maintenance with secukinumab 300 mg s.c. every 4 weeks for an additional 48 weeks.
  Interventions: Drug: Secukinumab 300mg s.c.
- Secukinumab 150 mg (Active Comparator): Induction with secukinumab 150 mg s.c. once per week (Week 0, 1, 2, 3 and 4) followed by maintenance with secukinumab 150 mg s.c. every 4 weeks for an additional 48 weeks.
  Interventions: Drug: Secukinumab 150mg s.c.

INTERVENTIONS:
Drug: Secukinumab 300mg s.c. — Induction: 5 x 150 mg secukinumab s.c. weekly. Maintenance: 300 mg secukinumab s.c. every 4 weeks
  Other Names: AIN457; Cosentyx
  Arms: Secukinumab 300mg
Drug: Secukinumab 150mg s.c. — Induction: 5 x 150 mg secukinumab s.c. weekly. Maintenance: 150 mg secukinumab s.c. every 4 weeks
  Other Names: AIN457; Cosentyx
  Arms: Secukinumab 150 mg

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of secukinumab 300mg in Chinese adults participants with active ankylosing spondylitis (AS) who have had an inadequate response to at least 2 non-steroidal anti-inflammatory drugs (NSAIDs) or intolerance to or a contraindication for NSAIDs, and who are naïve to biologic disease-modifying anti-rheumatic drugs (bDMARD).

DETAILED DESCRIPTION:
This study includes two periods: a 16-week double-blind placebo-controlled period and a 52-week open-label long-term extension period.

Eligible participants were randomly assigned in a 1:1 ratio to receive secukinumab 300 mg or placebo for 16 weeks in Period 1.

Participants who completed Period 1 received secukinumab 300 mg for 36 weeks in the extension period.

ELIGIBILITY:
Inclusion Criteria:

* Participant with a clinical diagnosis of ankylosing spondylitis (AS) and meeting the modified New York criteria for AS.
* Participant must have baseline disease activity as defined by having a Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) score >= 4 and a Patient's Assessment of ●Total Back Pain score >= 4 based on a 0 - 10 numeric rating scale (NRS) at the Screening and Baseline visits.
* Participant has had an inadequate response to at least two nonsteroidal anti-inflammatory drugs (NSAIDs) over an at least 4-week period in total at maximum recommended or tolerated doses, or participant has an intolerance to or contraindication for NSAIDs as defined by the Investigator.
* If entering the study on concomitant methotrexate (MTX), leflunomide, sulfasalazine (SSZ), and/or hydroxychloroquine, participant must be on a stable dose of MTX (<= 25 mg/week) and/or SSZ (<= 3 g/day) and/or hydroxychloroquine (<= 400 mg/day) or leflunomide (<= 20 mg/day) for at least 28 days prior to the Baseline visit. A combination of up to two background conventional synthetic disease-modifying anti-rheumatic drugs (csDMARDs) is allowed except the combination of MTX and leflunomide.
* If entering the study on concomitant oral corticosteroids, participant must be on a stable dose of prednisone (<= 10 mg/day), or oral corticosteroid equivalents, for at least 14 days prior to the Baseline visit.
* If entering the study on concomitant NSAIDs, tramadol, combination of acetaminophen and codeine or hydrocodone, and/or non-opioid analgesics, participant must be on stable dose(s) for at least 14 days prior to the Baseline visit.

Exclusion Criteria:

* Prior exposure to any Janus kinase (JAK) inhibitor (including but not limited to tofacitinib, baricitinib, and filgotinib).
* Prior exposure to any biologic therapy with a potential therapeutic impact on spondyloarthritis (SpA).
* Intra-articular joint injections, spinal/paraspinal injection(s), or parenteral administration of corticosteroids within 28 days prior to the Baseline visit. Inhaled or topical corticosteroids are allowed.
* Participant on any other DMARDs (other than those allowed), thalidomide or apremilast within 28 days or five half-lives (whichever is longer) of the drug prior to the Baseline visit.
* Participant on opioid analgesics (except for combination acetaminophen/codeine or acetaminophen/hydrocodone which are allowed) or use of inhaled marijuana within 14 days prior to the Baseline visit.
* Participant has a history of inflammatory arthritis of different etiology other than axial SpA (including but not limited to rheumatoid arthritis, psoriatic arthritis, mixed connective tissue disease, systemic lupus erythematosus, reactive arthritis, scleroderma, polymyositis, dermatomyositis, fibromyalgia), or any arthritis with onset prior to 17 years of age.
* Laboratory values meeting the following criteria within the Screening period prior to the first dose of study drug: serum aspartate transaminase > 2 × upper limit of normal (ULN); serum alanine transaminase > 2 × ULN; estimated glomerular filtration rate by simplified 4-variable Modification of Diet in Renal Disease formula < 40 milliliter (mL)/minute/1.73m^2; hemoglobin < 10 gram/deciliter, total white blood cell count < 2,500/microliter (μL); absolute neutrophil count < 1,500/μL; absolute lymphocyte count < 800/μL; and platelet count < 100,000/μL.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2024-06-14 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Assessment of SpondyloArthritis International Society (ASAS) 40 Response at Week 24 | 24 weeks
  ASAS 40 response was defined as improvement of ≥ 40% relative to Baseline and absolute improvement of ≥ 2 units (on a scale from 0 to 10) in ≥ 3 of the following 4 domains with no deterioration (defined as a net worsening of > 0 units) in the potential remaining domain:
  Patient's global assessment of disease activity, measured on a numeric rating scale (NRS) from 0 (no activity) to 10 (severe activity); Pain, measured by the total back pain NRS from 0 (no pain) to 10 (most severe pain); Function, measured by the Bath Ankylosing Spondylitis Functional Index (BASFI) which consists of 10 items assessing participants' ability to perform activities on an NRS ranging from 0 (easy) to 10 (impossible); Inflammation, measured by the mean of the 2 morning stiffness-related Bath AS Disease Activity Index (BASDAI) NRS scores (items 5 [level of stiffness] and 6 [duration of stiffness]) each on a scale from 0 (none/0 hours) to 10 (very severe/2 hours or more duration).

SECONDARY OUTCOMES:
Change From Baseline in Ankylosing Spondylitis Disease Activity Score (ASDAS) at Week 48 | Baseline and Week 48
  ASDAS is a composite index to assess disease activity in Ankylosing Spondylitis. ASDAS combines the following 5 disease activity variables using a weighted formula:
  Patient's assessment of total back pain (BASDAI Question 2; NRS score 0 [none] - 10 [very severe]) Patient global assessment of disease activity (NRS score 0 [no activity] - 10 [severe activity]) Peripheral pain/swelling (BASDAI Question 3; NRS score 0 [none] - 10 [very severe]) Duration of morning stiffness (BASDAI Question 6; NRS score 0 [0 hours] - 10 [2 or more hours]) High-sensitivity C-reactive protein (hs-CRP) in mg/L. The overall score ranges from 0 with no defined upper score; published ranges for disease activity states as defined by the ASDAS include Inactive disease (ASDAS < 1.3) and very high disease (ASDAS > 3.5). A negative change from Baseline score indicates improvement in disease activity.
Change From Baseline in Spondyloarthritis Research Consortium of Canada (SPARCC) Magnetic Resonance Imaging (MRI) Score for the Spine at Week 48 | Baseline and Week 48
  In the SPARCC MRI assessment of the spine, the entire spine is evaluated for active inflammation (bone marrow edema). Six discovertebral units (DVU) representing the 6 most abnormal DVUs were selected to calculate the MRI Spine SPARCC score. For each of the 6 DVUs, 3 consecutive sagittal slices were assessed in 4 quadrants to evaluate the extent of inflammation in all three dimensions.
  Each quadrant was scored for the presence (1) or absence (0) of edema. If edema was present in at least one quadrant of a DVU slice, it was also scored for intensity and depth of the edema representing that slice: An additional score of 1 was assigned if an intense signal was seen in any quadrant on a DVU slice. Slices that included a lesion demonstrating continuous increased signal of depth ≥ 1 cm extending from the endplate were scored as an additional 1 per slice.
  The maximum (worst) overall score for all 6 DVUs is 108.
Percentage of Participants With Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) 50 Response at Week 48 | Baseline and Week 48
  The BASDAI assesses disease activity by asking the participant to answer 6 questions (each on an 11 point numeric rating scale [NRS]) pertaining to symptoms experienced for the past week. For Questions 1 to 5 (level of fatigue/tiredness, level of AS neck, back or hip pain, level of pain/swelling in joints, other than neck, back or hips, level of discomfort from any areas tender to touch or pressure, and level of morning stiffness), the response is from 0 (none) to 10 (very severe); for Question 6 (duration of morning stiffness), the response is from 0 (0 hours) to 10 (≥ 2 hours). The overall BASDAI score ranges from 0 to 10. Lower scores indicate less disease activity.
  A BASDAI 50 response is defined as improvement of 50% or more from Baseline in BASDAI score.
Change From Baseline in Ankylosing Spondylitis Quality of Life (ASQoL) Score | Baseline and Week 48
  The ASQoL consists of 18 items related to quality of life, including the impact of pain on sleep, mood, motivation, ability to cope, activities of daily living, independence, relationships, and social life. Each item is answered as yes (scored as 1) or no (scored as 0).
  Scores are summed to obtain the overall score which ranges from 0 to 18, where higher scores indicate a worse quality of life. A negative change from Baseline in ASQoL indicates improvement in quality of life.
Percentage of Participants Achieving an Assessment of Spondyloarthritis International Society (ASAS) Partial Remission | Baseline and Week 48
  ASAS partial remission (PR) is defined as an absolute score of ≤ 2 units on a 0 to 10 scale for each of the four following domains:
  Patient's global assessment of disease activity, measured on a numeric rating scale (NRS) from 0 (no activity) to 10 (severe activity); Pain, measured by the total back pain NRS from 0 (no pain) to 10 (most severe pain); Function, measured by the Bath Ankylosing Spondylitis Functional Index (BASFI) which consists of 10 items assessing participants' ability to perform activities on an NRS ranging from 0 (easy) to 10 (impossible); Inflammation, measured by the mean of the 2 morning stiffness-related Bath AS Disease Activity Index (BASDAI) NRS scores (items 5 [level of stiffness] and 6 [duration of stiffness]) each on a scale from 0 (none/0 hours) to 10 (very severe/2 hours or more duration).
Change From Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) at Week 48 | Baseline and Week 48
  The Bath Ankylosing Spondylitis Functional Index is a validated index to determine the degree of functional limitation in patients with AS. BASFI consists of 10 questions assessing participants' ability to perform activities such as putting on socks, bending, reaching, getting up from the floor or an armless chair, standing, climbing and other physical activities. Each item is scored on a NRS ranging from 0 (easy to perform an activity) to 10 (impossible to perform an activity). The overall score is the mean of the 10 items and ranges from 0 to 10 with higher scores indicating more functional limitations. A negative change from Baseline in BASFI indicates improvement.
Change From Baseline in Linear Bath Ankylosing Spondylitis Metrology Index (BASMI[Lin]) at Week 48 | Baseline and Week 48
  The BASMI is a composite score based on 5 direct measurements of spinal mobility:
  cervical rotation (measured in degrees), tragus to wall distance (in centimeters [cm]) lumbar side flexion (in cm), lumbar flexion (modified Schober's) (in cm) and intermalleolar distance (in cm). Each measurement is converted to a linear score between 0 and 10. The total BASMI score is the average of the 5 scores and ranges from 0 to 10; the higher the BASMI score the more severe the patient's limitation of movement due to their ankylosing spondylitis. A negative change from Baseline indicates improvement.
Change From Baseline in Maastricht Ankylosing Spondylitis Enthesitis Score (MASES) at Week 48 | Baseline and Week 48
  The MASES evaluation was conducted to assess the presence or absence of enthesitis (inflammation of the entheses, or sites where tendons or ligaments insert into the bone) at 13 different sites (first costochondral joint left/right, seventh costochondral joint left/right, posterior superior iliac spine left/right, anterior superior iliac spine left/right, iliac crest left/right, fifth lumbar spinous process, and proximal insertion of Achilles tendon left/right. Each site was scored for presence (1) or absence (0) of enthesitis. The MASES is the sum of the 13 site scores, and ranges from 0 to 13, with higher scores indicating more inflammation of the entheses.
Change From Baseline in Work Productivity and Activity Impairment (WPAI) Overall Work Impairment at Week 48 | Baseline and Week 48
  The Work Productivity and Activity Impairment Questionnaire: Axial Spondyloarthritis, Version 2.0 (WPAI-Axial Spondyloarthritis) measures the effect of overall health and specific symptoms on productivity at work and outside of work. It consists of 6 questions. Respondents were asked about time missed from work and time while at work during which productivity was impaired in the past seven days. Results of WPAI are expressed as a percentage of impairment from 0 to 100, with higher percentages indicating greater impairment and less productivity. Overall Work Impairment indicates the percentage of overall work impairment due to health problems. A negative change from Baseline indicates improvement.
Change From Baseline in ASAS Health Index (HI) at Week 48 | Baseline and Week 48
  The ASAS HI measures functioning and health across 17 aspects of health in patients with AS, including pain, emotional functions, sleep, sexual function, mobility, self care, and community life. Each of the 17 questions is answered by the participant as "I agree" (score = 1) or "I disagree" (score = 0). The responses to the 17 dichotomous items are summed up to give a total score ranging from 0 to 17, where a higher score indicates a worse health status. A negative change from Baseline indicates improvement.
Percentage of Participants Achieving an ASAS 20 Response at Week 48 | Baseline and Week 48
  ASAS 20 response was defined as an improvement of ≥ 20% and an absolute improvement of ≥ 1 unit (on a scale of 0 to 10) from Baseline in at least 3 of the following 4 domains, with no deterioration (defined as a worsening of ≥ 20% and a net worsening of ≥ 1 units [on a scale of 0 to 10]) in the remaining domain:
  Patient's global assessment of disease activity, measured on a NRS from 0 (no activity) to 10 (severe activity); Pain, measured by the total back pain NRS from 0 (no pain) to 10 (most severe pain); Function, measured by the BASFI which consists of 10 items assessing participants' ability to perform activities on an NRS ranging from 0 (easy) to 10 (impossible); Inflammation, measured by the mean of the 2 morning stiffness-related BASDAI NRS scores (items 5 [level of stiffness] and 6 [duration of stiffness]) each on a scale from 0 (none/0 hours) to 10 (very severe/2 hours or more duration).
Change From Baseline in SPARCC MRI Score for Sacroiliac Joints at Week 48 | Baseline and Week 48
  In the SPARCC MRI assessment of the sacroiliac (SI) joints 6 consecutive sacroiliac joint image coronal slices representing the largest proportion of the synovial compartment of the SI joints were assessed for edema, intensity and depth of edema.
  Each SI joint (left and right) was divided into quadrants for a total of 8 SI scoring locations. Each quadrant was scored for the presence (1) or absence (0) of edema, intensity of edema (a score of 1 was assigned for each SI joint (left and right) if an intense signal was seen in any quadrant of that joint for each slice), and a lesion was graded as deep (score of 1) if there was homogeneous and unequivocal increase in signal extending over a depth of at least 1 cm from the articular surface of the SI joint in any quadrant.
  The total maximum score for all SI joints across 6 slices is 72.

CONTACTS AND LOCATIONS:
Overall Officials: AIHUA DU, M.D, Study Chair — Tongji Hospital
Locations (2):
- China (2):
  - Department of RheumatologyTongji Hospital, Wuhan, Hubei
  - Tongji Hospital, Wuhan, Hubei

IPD SHARING:
Plan to Share IPD: No